CLINICAL TRIAL: NCT04873999
Title: Prospective, Open, Non-interventional Study to Assess the Ability of an Electrical Impedance Tomograph (PlumoVista 500) to Monitor Changes in Lung Ventilation Over Time in Mechanically Ventilated Children.
Brief Title: Prospective, Open, Non-interventional Study to Assess the Ability of an Electrical Impedance Tomograph (PlumoVista 500)
Acronym: PV500ped
Status: Completed | Type: Observational
Sponsor: Drägerwerk AG & Co. KGaA (Industry)
Responsible Party: Sponsor
Other Study IDs: PV500ped
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Monitoring of Regional Distribution of Ventilation; Monitoring of Lung Volume

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational PMCF study will be conducted to generate and gather clinical data from the intended target population of pediatric patients.

The intention for Post-Market Clinical Follow-up (PMCF) is to confirm the performance and safety of a device throughout the device's lifecycle.

PulmoVista 500 is a lung function monitor for clinical use which continuously generates cross-sectional images of the lung function by applying the technique of electrical impedance tomography (EIT).

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric male or female patients excluding preterm infants
2. Patients with a chest circumference between 36 and 72 cm
3. Patients ≤ 12 years.
4. Patients with a tidal volume > 20 ml, i.e., children with a body weight of more than 3.3 kg (assuming a targeted tidal volume of 6 mL/kg body weight)
5. Patients for whom mechanical ventilation is intended
6. Patients whose regional distribution of ventilation and of lung volume are of clinical interest
7. Patients who are (should be) ventilated via an artificial airway access, whereby the ventilator used is compatible with PulmoVista 500
8. Patients and / or their legal guardians or legal representatives who have given written informed consent to participate in the study

Exclusion Criteria:

1. Patients who are supplied with a permanent or temporary pacemaker, an implantable defibrillator or other medical devices that emit electrical energy (e.g. cochlea amplifier implant)
2. Patients with a tidal volume ≤ 20 ml
3. Patients in whom the application of the electrode belt could be impaired by wound care or infections in the chest area
4. Female patients for whom pregnancy cannot be excluded; a pregnancy test should be performed at the discretion of the investigator.
5. Patients with an alleged allergic reaction to the materials of the electrode belt
6. Patients with a Body Mass Index (BMI) > 40
7. Evidence that suggests that the patient or their legal representative will not comply with the protocol requirements
8. Patients with a proven infectious disease (e.g. SARS-COV-19, MRSA) that requires isolation of the patient

Max Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric patients that visit the hospital for any kind of surgery, therefore requireing mechanical ventilation. Monitoring of Regional Distribution of Ventilation and Lung Volume are of clinical interest in these patients.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
assess the capability of PulmoVista 500 for continuous monitoring of ventilation | Duration per participant: 2 - 3 days (screening, procedure with PulmoVista 500, safety follow-up). Measurements with PulmoVista 500 per patient during mechanical ventilation is anticipated for a maximum of 10 minutes in total.
  To assess the capability of PulmoVista 500 for continuous monitoring of ventilation, the cross-correlation function (CCF) between the global impedance waveform of EIT and global tidal volume waveforms of a ventilator across multiple respiratory cycles in patients under controlled mechanical ventilation, will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Wolf, PD Dr., Principal Investigator — Children's hospital Traunstein
Locations (1):
- Klinik für Kinder- und Jugendmedizin Klinikum Traunstein, Traunstein, Germany

REFERENCES:
- [Derived] Clasen D, Winter I, Rietzler S, Wolf GK. Changes in ventilation distribution during general anesthesia measured with EIT in mechanically ventilated small children. BMC Anesthesiol. 2023 Apr 12;23(1):118. doi: 10.1186/s12871-023-02079-z. PMID 37046213